CLINICAL TRIAL: NCT05702281
Title: Evaluation of the Safety and Efficacy of the ReLARC Inserter During the Insertion Procedure of GYNEFIX Intrauterine Copper Bearing Contraceptive Device with a Follow-up of 3 Years.
Acronym: ReLARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REL-005
Record Dates: First submitted 2021-06-22; First posted 2023-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: copper intra-uterine device; Hysteroscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ReLARC 3 (Other): ReLARC® is a GyneFix® device intended to be inserted via hysteroscopy. Hysteroscopic insertion of the device allows direct visualization of the procedure, which makes it extremely safe.
  ReLARC® 3 is inserted through a hysteroscope (KARL STORZ HOPKINS® Wide Angle Straight Forward Telescope 6°, art. no. 26208AMA in combination with the irrigation pump Endomat® select).
  Interventions: Device: ReLARC
- ReLARC 10 (Other): ReLARC® is a GyneFix® device intended to be inserted via hysteroscopy. Hysteroscopic insertion of the device allows direct visualization of the procedure, which makes it extremely safe.
  ReLARC® 10 is inserted through a hysteroscope (KARL STORZ HOPKINS® Wide Angle Straight Forward Telescope 6°, art. no. 26208AMA in combination with the irrigation pump Endomat® select).
  Interventions: Device: ReLARC

INTERVENTIONS:
Device: ReLARC — ReLARC® is a GyneFix® device intended to be inserted via hysteroscopy. Hysteroscopic insertion of the device allows direct visualization of the procedure, which makes it extremely safe.

SUMMARY:
Insertion under vision such as hysteroscopy allows the ability to visualize the uterus prior to insertion, to assess uterine compatibility and the assurance of proper device placement. ReLARC® is a GyneFix® device intended to be inserted via hysteroscopy. Hysteroscopic insertion of the device allows direct visualization of the procedure, which makes it extremely safe.

This multicentre, open-label study will take place at the Women's Clinic of Ghent University Hospital in Belgium (International Coordinating Centre) and at the University Hospital AOU Federico II of Naples in Italy.

Primary aim:

To evaluate the safety of the ReLARC® inserter during the insertion procedure of GyneFix® intrauterine copper bearing contraceptive devices by means of successful placement with adequate position during follow-up evaluations.

Providing no complications develop, participants will remain in the study for 3 years. 120 women will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women, 18 - 48 years of age and not having a contraindication for hysteroscopy
* Be willing to come back for the follow-ups
* Be willing to refrain from having intercourse the first two weeks and using tampons and menstrual cups in the first 2 months, following insertion
* Sign a written informed consent
* Fundus thickness should be 11mm or more

Exclusion Criteria:

* T and Y shaped uterus
* U1, dysmorphic uterus (abnormal myometrium may result in bad device fixation)
* Complete septate U2b uterus
* Bicorporal U3-U6 uterus
* Injectables contraceptive use in the last 6 months
* The presence of infection of the uterus, clinical cervicitis or vaginitis (infection should be ruled out)
* Intrauterine fibroids (intra-mural, intracavitary or submucosal)
* Cancer or other disease of the uterus
* Malignancy, or treatment for malignancy. Melanoma or any gynaecological cancer at any time excludes the subject
* Blood clotting disorders
* Intrauterine polyps
* Subjects receiving corticosteroid therapy or immunosuppressive drugs
* Morbus Wilson
* AIDS
* Pregnancy

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Positioning of the ReLARC IUD | 3 years
  To evaluate the position of the ReLARC® IUD to confirm the succesful placement of the IUD with the ReLARC inserter during every follow-up visit.

SECONDARY OUTCOMES:
Ease of insertion | During Insertion visit
  1. The ease of the insertion (hysteroscope and ReLARC® device) by the following scale:
  1. Insertion went smoothly.
  2. I had little trouble while inserting the device but experienced this as a not important delay in my surgical act.
  3. Insertion was rather difficult.
  4. Insertion was time consuming, difficult, and dangerous.
  5. Insertion was not possible due to technical issues or medical reasons.
Learning curve of ReLARC insertion | During Insertion visit
  2. The learning curve of ReLARC® insertion, that starts after introducing the scope in the cervix and ends when the thread is cut and looped. This will be reported in minutes.
Pain score | During Insertion visit
  the participant's pain by a Visual Analogue Scale-VAS (1. no pain, 2. mild pain, 3. nasty pain, 4. severe pain, 5. unbearable pain) will be described.
patient satisfactory | 3 years after insertion
  The patient satisfactory score will be determined at every follow-up visit (4-8 weeks after insertion; 1 year after insertion, 2 years after insertion and 3 years after insertion)
Uterine cavity transverse diameter | During insertion visit
  the uterine cavity transverse diameter (UCTD) (before ReLARC® device insertion) will be described.
Expulsion rate | 7 years
  The number of expulsions of the IUD will be registered during the trial
Removal rate | 7 years
  The number of early removal of the IUD will be registered during the trial
Ease of removal | 7 years
  The ease of removal (Likert scale): 1. very easy, 2. easy, 3. neither easy nor difficult, 4. difficult, 5. very difficult
Pain at removal | 7 years
  pain (VAS): 1. no pain, 2. mild pain, 3. nasty pain, 4. severe pain, 5. unbearable pain

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No